CLINICAL TRIAL: NCT00125632
Title: Measuring Reading Rehabilitation Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: O3877R
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2006-12

CONDITIONS: Age Related Maculopathy; Retinal Degeneration
Keywords: Reading; Rehabilitation; Treatment Outcomes; Low vision
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Vision, Low

INTERVENTIONS:
Procedure: Eccentric Viewing Training for Reading

SUMMARY:
The purpose of this study is to measure the effectiveness of a newly-designed oculomotor training program for patients with age-related macular degeneration.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is currently among the top three leading causes of central vision loss in veterans (Chomsky et al., 1995) and is the most prevalent cause of blindness among veterans (37.2%, Quillen & Henry, 2000). The loss of central vision associated with these diseases has a profound impact on the quality of life of those affected, with many suffering depression. It is devastating to no longer be able to read a newspaper or recognize facial expressions. The use of preferred retinal locations (PRLs) to compensate for diseased foveae has offered hope to these patients in regaining some function. The investigators have developed a protocol that includes training in three major visual skills areas:

* visual awareness and eccentric viewing;
* reading eye movements; and
* processing of sequentially presented lexical information.

Module 1 focuses on making the patient aware of better vision at an eccentric location relative to degraded vision at the diseased fovea. Module 2 is focused on the improvement of the control of eye movements with the PRL. Module 3 is focused on reading practice without eye movements. These program curriculums and preliminary results are provided in the present proposal. The primary aim of this proposal is to quantitatively assess the relative effectiveness for improving reading and to establish the minimum training time need for skill improvement. Sixty patients with AMD who are already using a PRL will be selected to be similar in visual characteristics (e.g., visual acuity, contrast sensitivity, size of scotoma, duration of disease) and included in an experimental group. All patients in the experimental group will be trained with all three modules using a repeated measures - completely counterbalanced - design to control for training order effects. An additional 24 AMD patients will be recruited for a control group to be tested at the same time intervals as the experimental patients, but do not receive training between these assessment period intervals. The control group patients will be given the option to receive training following the assessment period. Both the experimental and the control patients will be assessed using the same outcome measures of reading (using MNRead Acuity Charts, the Pepper Visual Skills for Reading (VSR) Test, and the View Sentences Test). The performance of the experimental patients on the outcomes battery post-training will be compared to their pre-training performance on the same battery. Any change in performance of the experimental patients will be compared to the test-retest performance of the control patients. A questionnaire (the Veterans Administration Low Vision Visual Functioning Questionnaire) will also be administered to assess perceived abilities to perform everyday tasks before and following training. The control patients will also receive the questionnaire before and after their assessment period. In addition, the experimental patients will also be assessed on the exercises practiced during the module at the end of each daily training session to determine exactly when in the training protocol an improvement in performance on the exercises being trained has occurred. These daily performance measures provide for a finer scale for detecting performance changes. Statistical analyses will be conducted to answer the following key questions:

* What visual skills related to reading are trainable?
* Which methods are best for training these skills?
* What is the time course of visual skill improvement?
* Do the answers to these questions depend upon individual patient characteristics (e.g., age, disease severity, PRL location, cognitive factors)?
* Do patients who do not undergo training, but have repeated reading performance assessments, show improvements in reading skills?

Advances are being made in the area of retinal cell transplantation, gene therapy, and retinal prosthetics. When these techniques become part of standard clinical care, it is likely that the patients will require vision rehabilitation techniques to help them make sense of their potentially fragmented percepts. This research offers an evaluation of relative successes of the components of reading rehabilitation and will lead to the design of an efficient and effective composite training strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AMD
* An established preferred retinal locus
* Visual acuity of less than or equal to 20/70 and greater than or equal to 20/400 (in the better eye)

Exclusion Criteria:

* Those with other major ophthalmologic and neurologic disease; choroidal neovascularization ("wet" AMD); moderate to severe media opacities; and cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-08; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Participants will be given the following assessment tests at 4 different times during the assessment (at baseline, after 6 weeks, after 12 weeks, and after 18 weeks): eye tracking measures, daily performance measures and reading measures.

CONTACTS AND LOCATIONS:
Overall Officials: Janet P Szlyk, Ph.D., Principal Investigator — Research & Development Service 151, Jesse Brown VA Medical Center
Locations (1):
- Jesse Brown VA Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Szlyk JP, Paliga J, Seiple W, Rabb MF. Comprehensive functional vision assessment of patients with North Carolina macular dystrophy (MCDR1). Retina. 2005 Jun;25(4):489-97. doi: 10.1097/00006982-200506000-00015. PMID 15933597
- [Derived] Grant P, Seiple W, Szlyk JP. Effect of depression on actual and perceived effects of reading rehabilitation for people with central vision loss. J Rehabil Res Dev. 2011;48(9):1101-8. doi: 10.1682/jrrd.2010.05.0080. PMID 22234714
- [Derived] Seiple W, Grant P, Szlyk JP. Reading rehabilitation of individuals with AMD: relative effectiveness of training approaches. Invest Ophthalmol Vis Sci. 2011 May 5;52(6):2938-44. doi: 10.1167/iovs.10-6137. PMID 21296824
- See also: Related Info — http://www.uic.edu/com/eye/Research/Labs/lowvision/main.htm